CLINICAL TRIAL: NCT05299372
Title: Optimising the Management of Ventilated Patients and Quality of Life in Motor Neurone Disease: a Pilot Study
Brief Title: Telemonitoring in NIV MND (OptNIVent)
Acronym: OptNIVent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 767/14
Record Dates: First submitted 2021-09-21; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: non-invasive ventilation; Telehealth; Telemonitoring
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring via Careportal® (Other): Participants will be prompted by the device to answer two sets of questions every week: 10 items (1 nested) in the morning and 16 items (4 nested) in the evening. Also on a weekly basis, patients will be prompted to perform overnight oximetry test, and upload patient-ventilator interaction data (PVI) via Careportal®.
  Interventions: Other: Telemonitoring via Careportal®

INTERVENTIONS:
Other: Telemonitoring via Careportal® — The question sets and overnight oximetry results will be monitored and screened by a call centre commissioned by the Liverpool Clinical Commissioning Group (LCCG). The call centre will screen the weekly data and contact clinicians where appropriate (i.e. NIV team, MND specialist nurse, or patient's GP). PVI data will be examined by NIV physiotherapists, where required, following the contact from LCCG to ensure the maximum benefits of NIV to patients.

SUMMARY:
This is a feasibility study of telemonitoring system for people with MND/ALS, who are on NIV, via a call centre operated by a local clinical commissioning group.

DETAILED DESCRIPTION:
This study will test the feasibility of previously developed Telehealth system, using a device called Careportal®, to monitor people with MND/ALS who are using non-invasive ventilation (NIV). The Careportal® is a CE marked portable tablet computer device allowing telecommunication between patients and their care team through bespoke question sets, overnight oximetry test, and patient-ventilator interaction(PVI) data. Previously, the weekly telemonitoring via Careportal® was found to be an effective method to monitor symptom changes, allowing clinicians to optimise the care of ventilated patients with MND. This study will assess the practicality of using Careportal® in the care of ventilated patients with MND by monitoring patients through a patient support call centre. The call centre will screen the data and liaise with appropriate clinicians regarding changes of symptoms.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Confirmed diagnosis of MND with respiratory muscle weakness
* Adults who are capable of informed consent
* Patients for whom we anticipate survival of 6 months or more
* Able to communicate with an interviewer. Alternative communication methods will be used as required in order to mitigate communication difficulties.

Exclusion Criteria (Patients):

* Patients who have declined NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability - Qualitative data through semi-structured interviews and focus groups | Qualitative data will be conducted at 3-month
  Qualitative data will be collected through focus groups with participants, their lay caregivers, and clinicians. Separate focus groups will be conducted for the three participant groups with an option of individual interviews for patients and lay caregivers.
Usability - Qualitative data through semi-structured interviews and focus groups | Qualitative data will be conducted at 3-month
  Qualitative data will be collected through focus groups with participants, their lay caregivers, and clinicians. Separate focus groups will be conducted for the three participant groups with an option of individual interviews for patients and lay caregivers.

SECONDARY OUTCOMES:
Patient Reported Outcome Measurement - Neurological Fatigue Index for MND | Baseline and then 6-weekly up to 24 weeks
  13-item questionnaire assessing fatigue experienced by people with motor neurone disease. The questionnaire consists of two sub-scales: Weakness sub-scale and Energy sub-scale. Eight items make up the Summary Fatigue scale with the total scores range from 0 to 24. Higher scores indicate higher levels of fatigue
Patient Reported Outcome Measurement - Epworth Sleepiness Scale | Baseline and then 6-weekly up to 24 weeks
  8-item questionnaire to measure general levels of sleepiness. Total scores range from 0 to 24. Higher scores indicate higher levels of sleepiness.
Patient Reported Outcome Measurement - Dyspnoea-12 | Baseline and then 6-weekly up to 24 weeks
  12-item questionnaire to measure overall breathlessness severity. Total scores range from 0 to 36. Higher scores indicate higher breathless severity.
Patient Reported Outcome Measurement - revised Amyotrophic Lateral Sclerosis Functional Rating Scale | Baseline and at 3-month and 6-month
  12-item questionnaire to monitor the disease progression covering bulbar, motor and respiratory function. Total scores range from 0 to 48. Higher scores indicate better function.
Patient Reported Outcome Measurement - Hospital Anxiety and Depression Scale | Baseline and at 3-month and 6-month
  14-item questionnaire to measure anxiety and depression levels. The questionnaire consists of anxiety sub-scale and depression sub-scale. Scores for each sub-scale range from 0 to 21. Higher scores indicate greater anxiety/depression levels.
Patient Reported Outcome Measurement - the World Health Organization Quality of Life Scale-BREF | Baseline and at 3-month and 6-month
  26-item questionnaire consists of Physical Health domain, Psychological domain, Social relationships domain, and Environment domain in addition to Overall QoL (1-item) and General Health (1-item) facets. Total scores range from 0 to 100. Higher scores indicate indicate higher quality of life.
Patient Reported Outcome Measurement - 5-level EQ-5D | Baseline and at 3-month and 6-month
  The questionnaire consists of 5-item to measure health based on five domains: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each domain has 5 levels indicating worsening health, from having no problems to having severe problems. The questionnaire also contain one visual analogue scale measuring health-reported health: 0 indicates worst health while 100 indicates the best health.
Patient Reported Outcome Measurement - General Satisfaction | Baseline and at 3-month and 6-month
  6-item General Satisfaction sub-scale from Patient Satisfaction Questionnaire. Total scores range from 6 to 30. Higher scores indicate greater satisfaction.
Patient Reported Outcome Measurement - Access, Availability and Convenience | Baseline and at 3-month and 6-month
  12-item Access, Availability and Convenience sub-scale from Patient Satisfaction Questionnaire. Total scores range from 12 to 60. Higher scores indicate greater access, availability and convenience.
Self-Reported Outcome Measurement - Caregiving Distress Scale | Baseline and at 3-month and 6-month
  17-item questionnaire to measure caregiver distress, covering five dimensions: Relationship distress, Emotional burden, Social impact, Care-receiver demands, and Personal cost. Total scores range from 0 to 68. Higher scores indicate greater distress.
Service evaluation | At the end of study i.e. at 6-month
  Patient Level Information and Costing System (PLICS)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Angus, MRCP, FRCP, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust

REFERENCES:
- [Background] Ando H, Ashcroft-Kelso H, Halhead R, Young CA, Chakrabarti B, Levene P, Cousins R, Angus RM. Incorporating self-reported questions for telemonitoring to optimize care of patients with MND on noninvasive ventilation (MND OptNIVent). Amyotroph Lateral Scler Frontotemporal Degener. 2019 Aug;20(5-6):336-347. doi: 10.1080/21678421.2019.1587630. Epub 2019 Mar 26. PMID 30912468